CLINICAL TRIAL: NCT01739010
Title: Efficacy of Intravenously Instituted Hypothermia Treatment in Improving Functional Outcomes in Patients Following Acute Spinal Cord Injury
Brief Title: Hypothermia Following Acute Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Allan D. Levi, MD, PhD, Professor of Neurosurgery, University of Miami
Other Study IDs: 20060556
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate the long term outcome of patients who receive hypothermia treatment for spinal cord injury. At this institution, intravascular hypothermia has been used for certain patients with spinal cord injury for the past two years. This study will collect data from vital signs and examinations while the patient is in the hospital and also when they follow up as an outpatient after they are discharged or go to a rehabilitation center. This data will then be analyzed and compared only to historically published data from previous studies. The aim of this investigation is to determine if intravascular hypothermia results in a beneficial outcome for patients with spinal cord injury.

DETAILED DESCRIPTION:
It is standard practice at this institution for patients with complete acute spinal cord injury to receive hypothermia. Incomplete injuries may also be treated with hypothermia. This will be a prospective analysis of the data collected at our institution from patients with acute spinal cord injury receiving the hypothermia protocol. The care of these patients will not be affected by this research. Data for normothermia (37 degrees Celsius) will be obtained from historical studies analyzing similar patient groups. Patients arriving to this emergency department have a baseline neurological examination in a timely fashion prior to the induction of hypothermia by a neurosurgical attending or resident. All patients have Magnetic Resonance Imaging (MRI) of the injured spinal cord on admission. Patients that are intubated and medically sedated prior to the initial exam by the neurosurgical team are excluded because the exam at that time may be inaccurate. Patients receiving hypothermia are transferred to the Neurosurgical ICU, intubated and sedated using muscle relaxants. Additional forms of sedation including benzodiazepines or dexmedetomidine are routinely used as an adjunct to curtail a shivering response. For all patients receiving hypothermia, an Alsius CoolGard® Icy Catheter is placed into the Inferior Vena Cava (IVC) via the femoral vein and the temperature cooled to target (33 degrees) at the maximum rate (0.5 degrees/hr). Mean arterial pressure (MAP) is kept >90 mm Hg at all times with fluid boluses (Normal Saline or Albumin 5%) or blood transfusions to keep the hematocrit at 30. Hypothermia at 33 degrees is maintained for 48 hours. Blood cultures are performed daily (from both a peripheral site and from the catheter itself) and an Orogastric tube (OGT) or Nasogastric tube (NGT) is placed in each patient. Nutrition is provided as per our current nutritional supplementation protocol. Intravenous fluids consist of Normal Saline at all times unless the serum Na rises above 160. Serum electrolytes, coagulation studies and complete blood count are performed daily. After 48 hours of hypothermia, the patient is rewarmed to 37 degrees at a controlled rate of 0.1 degree/hr. After reaching 37 degrees, the intravenous catheter is maintained for no more than 6 days total to keep the systemic temperature at 37 degrees. Surface cooling techniques are occasionally utilized for the purpose of maintaining normothermia after 6 days. The patients are discharged to rehabilitation after they are stabilized. All patients will be reevaluated at 6 weeks, 6, and 12 months using the American Spinal Injury Association (ASIA) sensory and motor scales with Functional Independence Measures (FIM). A follow-up MRI scan will be done at one year.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years of age, ASIA (American Spinal Injury Association) Impairment Scale (AIS) Score A or B, non-penetrating injury, and absence of severe systemic injury or coagulopathy. Patients urgently taken to the OR for reduction may also be included.

Exclusion Criteria:

* Age > 65 years, ASIA (American Spinal Injury Association) Impairment Scale (AIS) Score C or D, Hyperthermia on admission (> 37 degrees Celsius), Severe systemic injury, Severe bleeding, Pregnancy, Coagulopathy, Thrombocytopenia, Known prior cardiac history, Blood dyscrasia, Pancreatitis, Raynuad's syndrome, Penetrating spinal column injury (gunshot and knife wounds etc.), Cord transection. Patients who are intubated and sedated prior to initial examination by the neurosurgical team and patients showing an improvement in the neurologic exam within 12 hours from the injury will also be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute spinal cord injury patients.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
International Standards of Neurological Classification for Spinal Cord Injury | Change from Baseline at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Allan D Levi, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- Jackson Memorial Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No